CLINICAL TRIAL: NCT05658900
Title: Three-dimensional Volumetric Analysis of Bone Regeneration Following Jaw Cysts Enucleation With and Without Autologous Albumin Gel-platelet-rich Fibrin Mixture (A Randomized Controlled Clinical Trial)
Brief Title: Volumetric Analysis of Bone Following Jaw Cysts Enucleation With and Without Alb-PRF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cysts_2022
Record Dates: First submitted 2022-12-12; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Jaw Cysts
MeSH Terms: conditions — Jaw Cysts

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enucleation with albumin PRF (Experimental)
  Interventions: Other: Enucleation with albumin PRF
- Enucleation without albumin PRF (Active Comparator)
  Interventions: Other: Enucleation without albumin PRF

INTERVENTIONS:
Other: Enucleation with albumin PRF — The protocol that will be used in the preparation of albumin PRF
  1. A sample of venous blood, at ten milliliters, at least will be drawn from the patient in a sterile centrifuge tube.
  2. The venous blood sample will be centrifuged at 700 g for 8 minutes.
     * Betadine: Povidone-iodine, 7.5% (0.75% available iodine), Purdue Products L.P
  3. The platelet-poor plasma layer will be taken and heated at uniform temperature 75 celsius for 10 minutes in a thermostatic water bath incubator to denature albumin protein forming albumin gel.
  4. Once the albumin gel is cooled, to room temperature for 10 minutes, it will be mixed with the buffy coat layer of PRF using 3 way stop cock and 2 plastic syringes with Luer lock to obtain albumin PRF then leave it in the dappen dish for 5 minutes.
  Arms: Enucleation with albumin PRF
Other: Enucleation without albumin PRF — The full-thickness mucoperiosteal flap will be performed using blade no. 15 and Bard- Parker handles extending one tooth anterior and one tooth posterior to the cystic cavity.
  The mucoperiosteal flap will be reflected using the periosteal elevator to expose the bone.
  Removal of the overlying bone to expose the cystic lesion. Enucleation of the cyst.
  Arms: Enucleation without albumin PRF

SUMMARY:
Cyst is the main cause for longstanding swelling in the mandible or the maxilla, its enlargement usually results in resorption and weakening of bone. Thus the treatment of the cysts is essential to preserve the bone and the adjacent vital structures. Healing of the bone defect and its surrounding soft tissues is a critical issue that needs concerns. Although the Platelet rich fibrin has promising effects in wound healing, it can resorb during 10-14 days. Thus a new autologous platelet concentrate is introduced by Kawasi et al that can remain stable for 4-6 months called albumin PRF.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from jaw cystic cavity volume greater than 1cm3
* Patients with no gender predilection that agreed to present for follow-up visits for a minimum postoperative period of 6 months.
* Cystic lesion that requires removal under local or general anaesthesia.

Exclusion Criteria:

* Medically compromised patients contradicting operation.
* Patients with history of chemotherapy or radiotherapy.
* Patients with low level of platelet count.
* Patients with anticoagulant therapy.
* Patients who are unable to attend follow up appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2023-03-09 (Estimated); Study Completion 2023-03-09 (Estimated)

PRIMARY OUTCOMES:
Change in pain score | Up to 1 week
  It will be assessed on 3rd and 7th day through a 10-point Visual Analogue Scale (VAS)(25) (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe)
Change in soft tissue healing | up to 2 weeks
  it will be used using Landry index Healing Index 1: Very poor (has two or more of the following) Healing Index 2: Poor Healing Index 3: Good Healing Index 4: Very good Healing Index 5: Excellent
change in bone volume | at baseline and 6 months
  it will be assessed using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt

REFERENCES:
- [Derived] Shokry MMEM, Melek LNF, Amer TA. Three-dimensional volumetric analysis of bone regeneration following jaw cyst enucleation with and without an autologous albumin gel-platelet-rich fibrin mixture (Alb-PRF): a randomized controlled clinical trial. BMC Oral Health. 2025 May 8;25(1):693. doi: 10.1186/s12903-025-06027-w. PMID 40340767